CLINICAL TRIAL: NCT07396558
Title: Efficacy of Intermittent Erector Spinae Plane Block Via Subcutaneous Port for Cancer-Related Pain in Patients With Lung Cancer
Brief Title: Intermittent Erector Spinae Plane Block Via Subcutaneous Port for Cancer Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESPB_HMU2628
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Cancer Pain; Erector Spinae Plane Block
Keywords: Erector Spinae Plane Block; Regional Anesthesia; Cancer-Related Pain; Lung Cancer; Subcutaneous Port; Palliative Care
MeSH Terms: conditions — Cancer Pain; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design including an intervention group receiving intermittent erector spinae plane block via a subcutaneous port and a historical control group consisting of patients who received standard pain management prior to the implementation of the intervention. Outcomes are compared between the intervention group and the historical control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block Group (Experimental): Patients receive intermittent erector spinae plane block administered via a subcutaneous port as part of multimodal pain management for cancer-related pain.
  Interventions: Procedure: Erector Spinae Plane Block
- Historical Control Group (No Intervention): Historical control group consisting of patients with lung cancer who previously received standard pain management without erector spinae plane block.

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Intermittent erector spinae plane block administered via a subcutaneous port, allowing repeated delivery of local anesthetic for the management of cancer-related pain in patients with lung cancer.
  Arms: ESP Block Group

SUMMARY:
Cancer-related pain is a common and challenging problem in patients with lung cancer, often requiring long-term pain management. Conventional pain treatments, including systemic medications, may not provide adequate relief or may cause significant side effects.

The erector spinae plane (ESP) block is a regional anesthesia technique that can help reduce pain by delivering local anesthetic near the nerves supplying the chest wall. This study aims to evaluate the effectiveness and safety of intermittent ESP block administered through a subcutaneous port for controlling cancer-related pain in patients with lung cancer.

Eligible patients with lung cancer and moderate to severe pain will receive intermittent ESP block injections via a subcutaneous port as part of their pain management plan. Pain intensity, analgesic requirements, and potential side effects will be assessed over time.

The results of this study may help determine whether intermittent ESP block via a subcutaneous port is a useful and feasible option for improving pain control and quality of life in patients with lung cancer.

DETAILED DESCRIPTION:
Cancer-related pain in patients with lung cancer is often multifactorial and may be difficult to control using conventional systemic analgesic therapies alone. Regional anesthesia techniques have increasingly been explored as adjunctive approaches to improve pain control while minimizing systemic opioid exposure.

The erector spinae plane (ESP) block is a fascial plane block in which local anesthetic is injected adjacent to the erector spinae muscle, allowing spread to the dorsal and ventral rami of spinal nerves. This technique has been reported to provide effective analgesia for thoracic and chest wall pain with a favorable safety profile.

In this study, patients with lung cancer experiencing moderate to severe cancer-related pain will receive intermittent ESP block administered through a subcutaneous port. The port system allows repeated administration of local anesthetic without the need for repeated needle insertion, potentially improving patient comfort and feasibility of long-term pain management.

Pain intensity will be assessed using standardized pain assessment tools at predefined time points. Additional outcomes include changes in analgesic medication requirements, patient-reported comfort, and the occurrence of procedure-related or treatment-related adverse events.

This study is designed to evaluate the feasibility, effectiveness, and safety of intermittent ESP block via a subcutaneous port as part of a multimodal pain management strategy in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria

* Adult patients diagnosed with advanced-stage lung cancer who are currently receiving palliative care only.
* Presence of chronic cancer-related chest pain lasting longer than 1 month, localized to the thoracic region due to chest wall invasion, pleural involvement, or bone metastases.
* Performance status ≤ 3 according to the Eastern Cooperative Oncology Group (ECOG), allowing placement of a subcutaneous port and maintenance of local anesthetic administration.
* Inadequate pain control with conventional analgesic therapies or clinical indication for the addition of regional analgesia.
* Ability to understand the study procedures and provide written informed consent after receiving a full explanation of the intervention.

Exclusion Criteria:

* Chest pain with radiation to the upper extremities, neck, or shoulder, suggestive of non-localized thoracic pain.
* Severe hepatic or renal dysfunction, or severe heart failure (New York Heart Association class III-IV).
* Local infection at the injection or port placement site, or uncontrolled systemic infection.
* Severe cachexia or insufficient subcutaneous tissue that does not allow safe coverage of the subcutaneous port.
* Known allergy to amide-type local anesthetics or other contraindications to regional anesthesia.
* Severe cognitive impairment, altered consciousness, or inability to cooperate with post-intervention monitoring.
* Lack of adequate caregiver support for home-based follow-up after discharge or inability to coordinate follow-up with local healthcare facilities.
* Severe coagulation disorders, defined as:

  * International normalized ratio (INR) > 1.5
  * Activated partial thromboplastin time (aPTT) > 40 seconds
  * Fibrinogen < 1.5 g/L
  * Platelet count < 50 × 10⁹/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale (VAS) at Home at 3 Months After Discharge | From hospital discharge to 3 months after discharge
  Pain intensity is assessed at rest and during movement using a 10-cm Visual Analog Scale (VAS), where 0 represents no pain and 10 represents the worst imaginable pain. Assessments are performed at predefined home-based follow-up time points after hospital discharge.
  The primary outcome is the change in VAS pain score from hospital discharge to 3 months after discharge, reflecting the sustained effectiveness of intermittent erector spinae plane block in home-based palliative care. Outcomes in the intervention group will be compared with those of the historical control group.

SECONDARY OUTCOMES:
Change in Pain Intensity at Early Time Points After Intervention | From baseline (H0) to 30 minutes after intervention (H1) and at the time of transfer to the ward (H2)
  Pain intensity at rest and during movement is assessed using the Visual Analog Scale (VAS) at baseline, 30 minutes after the intervention, and at the time of transfer to the ward to evaluate the early analgesic effect of the erector spinae plane block.
Pain Intensity Trajectory During Home-Based Follow-Up | Pain intensity at rest and during movement is measured using the Visual Analog Scale (VAS) at predefined home-based follow-up time points up to 3 months after discharge to describe the trajectory of pain control during home-based palliative care.
  At predefined home-based follow-up time points on days 1, 3, and 5; weeks 1, 2, and 3; and months 1, 2, and 3 after hospital discharge
Morphine Consumption During Home-Based Palliative Care | At predefined home-based follow-up time points on days 1, 3, and 5; weeks 1, 2, and 3; and months 1, 2, and 3 after hospital discharge
  The daily dose of opioid analgesics used for rescue pain management during home-based follow-up is recorded and converted to morphine-equivalent doses to evaluate changes in opioid requirements over time.
Procedure-Related and Treatment-Related Adverse Events | At predefined home-based follow-up time points on days 1, 3, and 5; weeks 1, 2, and 3; and months 1, 2, and 3 after hospital discharge
  Procedure-related and treatment-related adverse events are recorded, including respiratory and hemodynamic changes after intervention, catheter-related complications, local anesthetic systemic toxicity, and opioid-related adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fallon M, Giusti R, Aielli F, Hoskin P, Rolke R, Sharma M, Ripamonti CI; ESMO Guidelines Committee. Management of cancer pain in adult patients: ESMO Clinical Practice Guidelines. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv166-iv191. doi: 10.1093/annonc/mdy152. No abstract available. PMID 30052758
- [Background] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016